CLINICAL TRIAL: NCT00195117
Title: A Randomized Trial of Changing Exercise and Physical Activity Behavior in Asthma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Mary E. Charlson, MD, Principal Investigator, Weill Medical College of Cornell University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: N01-HC-25196 (030200599); N01HC25196 (NIH)
Record Dates: First submitted 2005-09-14; First posted 2005-09-19 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Asthma
Keywords: Asthma; Behavior change; Physical activity; Risk reduction
MeSH Terms: conditions — Asthma; Motor Activity; Risk Reduction Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): This group received follow-up every 2-months for one year. Follow-up included questions about their asthma and how well they had been able to engage in their doctor approved physical activity goal.
- Intervention Group (Experimental): This group received follow-up every 2-months for one year. Follow-up included questions about their asthma and how well they had been able to engage in their doctor approved physical activity goal, which was the same as the control arm. Additionally, subjects in this arm were encouraged to use positive affect and self-affirmation techniques to motivate an increased level of participation in their physical activity goal. These subjects also received small token gifts to remind them of their participation in this study.
  Interventions: Behavioral: Intervention Group

INTERVENTIONS:
Behavioral: Intervention Group — Subjects were randomly assigned to either the control or the intervention group. The intervention included receiving an additional educational workbook about using positive affect and self affirmation, as well as participating in using positive affect and self-affirmation to motivate behavior change, which in this case was to increase their physical activity level. Patient also received small token gifts to remind them of their participation in the study and to induce positive affect. The control group also set a physical activity goal and received the same follow-up, but did not participate in the positive affect and self-affirmation portion.
  Other Names: Positive affect and self-affirmation induction
  Arms: Intervention Group

SUMMARY:
The primary objective of this randomized trial is to evaluate a novel intervention of induced positive affect and induced self-affirmation to increase physical activity in patients with asthma.

DETAILED DESCRIPTION:
The primary objective of this randomized trial is to evaluate a novel intervention of induced positive affect and induced self-affirmation to increase physical activity in patients with asthma. At the start of the trial all patients in conjunction with their physicians will select a program of mild to moderate physical activity or exercise to be adopted and maintained on a routine basis. All patients will record perceived exertion and pedometer measurements in a log diary. All patients will be contacted by telephone at set time intervals to encourage them to continue their selected physical activity or exercise. Patients randomized to the intervention arm will also receive induced positive affect and self-affirmation throughout the study period. Patients in the control arm will not receive the positive affect and self-affirmation components.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for this study

* if their physicians consider them medically able to participate, if they are 18 years of age or older
* if they have a diagnosis of mild to moderate asthma based on the NHLBI Asthma Expert Panel's classification system which rates symptoms, frequency of exacerbations, nocturnal attacks, activity restriction, use of medications, and pulmonary function.

Exclusion Criteria:

Patients will be excluded from this study for the following reasons:

* If they are unable to walk several blocks for whatever reason;
* If they have musculoskeletal or neurological deficits that preclude increased physical activity;
* If they have other pulmonary diseases;
* If they have cardiac disease or other severe comorbidity;
* If they are unable to provide informed consent because of cognitive deficits;
* If they refuse to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2004-10 (Actual); Primary Completion 2006-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be change in Paffenbarger Physical Activity and Exercise Index scores from enrollment to 12 months. | every 2 months for 1 year

SECONDARY OUTCOMES:
Pedometer readings from enrollment to 12 months. | every 2 months for 1 year
Change in asthma status measured by the Asthma Control Questionnaire from enrollment to 12 months. | baseline and one year after enrollment at closeout
Change in quality of life measured by the Asthma Quality of Life Questionnaire enrollment to 12 months. | at baseline, 4-,8-month follow-ups and one year after enrollment at closeout
Changes in the SF-12 from enrollment to 12 months. | baseline and one year after enrollment at closeout

CONTACTS AND LOCATIONS:
Overall Officials: Carol A Mancuso, MD, Principal Investigator — Weill Medical College of Cornell University; Mary E Charlson, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- New York Presbyterian Hospital-Weill Medical College of Cornell University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No Plan to Share IPD

REFERENCES:
- [Background] Mancuso CA, Peterson MG. Different methods to assess quality of life from multiple follow-ups in a longitudinal asthma study. J Clin Epidemiol. 2004 Jan;57(1):45-54. doi: 10.1016/S0895-4356(03)00248-8. PMID 15019010
- [Background] Mancuso CA, Rincon M, Robbins L, Charlson ME. Patients' expectations of asthma treatment. J Asthma. 2003 Dec;40(8):873-81. doi: 10.1081/jas-120023578. PMID 14736086
- [Background] Mancuso CA, Rincon M, McCulloch CE, Charlson ME. Self-efficacy, depressive symptoms, and patients' expectations predict outcomes in asthma. Med Care. 2001 Dec;39(12):1326-38. doi: 10.1097/00005650-200112000-00008. PMID 11717574
- [Background] Mancuso CA, Peterson MG, Charlson ME. Comparing discriminative validity between a disease-specific and a general health scale in patients with moderate asthma. J Clin Epidemiol. 2001 Mar;54(3):263-74. doi: 10.1016/s0895-4356(00)00307-3. PMID 11223324
- [Background] Mancuso CA, Peterson MG, Charlson ME. Effects of depressive symptoms on health-related quality of life in asthma patients. J Gen Intern Med. 2000 May;15(5):301-10. doi: 10.1046/j.1525-1497.2000.07006.x. PMID 10840265
- [Result] Mancuso CA, Choi TN, Westermann H, Wenderoth S, Hollenberg JP, Wells MT, Isen AM, Jobe JB, Allegrante JP, Charlson ME. Increasing physical activity in patients with asthma through positive affect and self-affirmation: a randomized trial. Arch Intern Med. 2012 Feb 27;172(4):337-43. doi: 10.1001/archinternmed.2011.1316. Epub 2012 Jan 23. PMID 22269593
- [Derived] Mancuso CA, Choi TN, Westermann H, Wenderoth S, Wells MT, Charlson ME. Improvement in asthma quality of life in patients enrolled in a prospective study to increase lifestyle physical activity. J Asthma. 2013 Feb;50(1):103-7. doi: 10.3109/02770903.2012.743150. Epub 2012 Nov 22. PMID 23173979
- [Derived] Mancuso CA, Sayles W, Allegrante JP. Development and testing of the Asthma Self-Management Questionnaire. Ann Allergy Asthma Immunol. 2009 Apr;102(4):294-302. doi: 10.1016/S1081-1206(10)60334-1. PMID 19441600
- [Derived] Westermann H, Choi TN, Briggs WM, Charlson ME, Mancuso CA. Obesity and exercise habits of asthmatic patients. Ann Allergy Asthma Immunol. 2008 Nov;101(5):488-94. doi: 10.1016/S1081-1206(10)60287-6. PMID 19055202
- [Derived] Choi TN, Westermann H, Sayles W, Mancuso CA, Charlson ME. Beliefs about asthma medications: patients perceive both benefits and drawbacks. J Asthma. 2008 Jun;45(5):409-14. doi: 10.1080/02770900801971834. PMID 18569235
- [Derived] Mancuso CA, Westermann H, Choi TN, Wenderoth S, Briggs WM, Charlson ME. Psychological and somatic symptoms in screening for depression in asthma patients. J Asthma. 2008 Apr;45(3):221-5. doi: 10.1080/02770900701883766. PMID 18415830
- [Derived] Mancuso CA, Wenderoth S, Westermann H, Choi TN, Briggs WM, Charlson ME. Patient-reported and physician-reported depressive conditions in relation to asthma severity and control. Chest. 2008 May;133(5):1142-8. doi: 10.1378/chest.07-2243. Epub 2008 Feb 8. PMID 18263683
- [Derived] Mancuso CA, Choi TN, Westermann H, Briggs WM, Wenderoth S, Charlson ME. Measuring physical activity in asthma patients: two-minute walk test, repeated chair rise test, and self-reported energy expenditure. J Asthma. 2007 May;44(4):333-40. doi: 10.1080/02770900701344413. PMID 17530534